CLINICAL TRIAL: NCT02637882
Title: The Effect of Applying Multidisciplinary Bundle Intervention on the Delirium Incidence in Critically Ill Patients
Acronym: Ghada
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Shalaby, principal investigator, Assiut University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Ghada 021
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Ear Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- First intervention (ear plug) (Experimental): Other: ear plug
  Other Name: eastnova ear plug
  Interventions: Other: Ear plug
- Second intervention (eye mask) (Other): Other: eye mask
  The patients will receive the second intervention (eye mask) in the second night (N2) from 9 pm to 6 am.
  Other Name: Sleeping mask
  Interventions: Other: Eye mask
- Ear plug and eye mask (Other): The patients will receive the mixed intervention (eye mask) and (ear plug ) in the first night (N1) from 9 pm to 6 am.
  Interventions: Other: Mixed intervention (ear plug and eye mask)

INTERVENTIONS:
Other: Ear plug — The patients will receive the first intervention (ear plug) in the third night (N3) from 9 pm to 6 am.and the patient will complete the sleep questionnaire sheet and delirium scale.
  Other Names: eastnova ear plug
  Arms: First intervention (ear plug)
Other: Eye mask — The patients will receive the second intervention (eye mask) in the second night (N2) from 9 pm to 6 am.and the patient will complete the sleep questionnaire sheet and delirium scale
  Other Names: Sleeping mask
  Arms: Second intervention (eye mask)
Other: Mixed intervention (ear plug and eye mask) — The patients will receive the intervention (eye mask and ear plug) in the first night (N1) from 9 pm to 6 am.and the patient will complete the sleep questionnaire sheet and delirium scale
  Other Names: ear plug and eye mask
  Arms: Ear plug and eye mask

SUMMARY:
The patients will exposed to different intervention through three nights (ear plug, eye mask). 50 patients in the age range 18- 60 years admitted to ICU of Assiut university hospitals will be randomly allocated into into two groups (control group and intervention group).

DETAILED DESCRIPTION:
The multicomponent bundle of interventions is designed to be multidisciplinary, and included measures taken to reduce noise, light and iatrogenic sleep disturbance, as well as attempts to modify risk factors for delirium. The patients will exposed to different intervention through three nights (ear plug, eye mask) grouping of nursing activity to be delivered before the 23:00 or delay their completion until after 08:00 where possible. Orientate patients regarding time, place and date every eight hours.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* No hearing problems.
* No eye disease.

Exclusion Criteria:

* Head injury.
* Psychiatric disease.
* Shocked patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-05 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
decrease delirium incidence | 8 month
  the patients will exposed to multi-component bundle

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Sh Khalaf, Lecturer, Principal Investigator — faculty of nursing ,Assuit university
Locations (1):
- Assuit university hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the patient's assessment sheet will be used to collect the data,the researcher will interview with the patient to complete the sleeping quality sleeping questionnaire and delirium scale

REFERENCES:
- [Background] Hellstrom A, Willman A. Promoting sleep by nursing interventions in health care settings: a systematic review. Worldviews Evid Based Nurs. 2011 Sep;8(3):128-42. doi: 10.1111/j.1741-6787.2010.00203.x. Epub 2010 Oct 12. PMID 21040451
- [Background] Dave K, Ashia Qureshi, L.Gopichandran, Usha Kiran. Effects of Earplugs and Eye Masks on Perceived Quality of Sleep during Night among Patients in Intensive Care Units. International Journal of Science and Research (IJSR) ISSN (Online): 2319-7064 Index Copernicus Value (2013): 6.14 | Impact Factor (2013): 4.438.
- [Background] Rivosecchi RM, Smithburger PL, Svec S, Campbell S, Kane-Gill SL. Nonpharmacological interventions to prevent delirium: an evidence-based systematic review. Crit Care Nurse. 2015 Feb;35(1):39-50; quiz 51. doi: 10.4037/ccn2015423. PMID 25639576